CLINICAL TRIAL: NCT00539253
Title: Assessment of Liver Cancer Response to Transcatheter Arterial Chemoembolization (TACE) Using Functional Triple-Phase MultiHance-Enhanced Magnetic Resonance Imaging (MRI)
Brief Title: Assessment of Liver Cancer Response to TACE Using MultiHance-Enhanced MRI.
Acronym: TACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J06108; NA_00003943 (Other: Johns Hopkins I.R.B.)
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — gadobenic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadobenate Dimeglumine (Multi Hance) (Other): If patient did not participate in this study (by signing consent), they could receive any other contrast used routinely at this facility including the contrast used in this study
  Interventions: Drug: gadobenate dimeglumine (MultiHance)

INTERVENTIONS:
Drug: gadobenate dimeglumine (MultiHance) — The contrast agent, gadobenate dimeglumine, will be used during MR imaging for both the baseline and 1 month f/u studies.
  Other Names: MultiHance

SUMMARY:
This research is being done to find out if using the contrast agent MultiHance can be used to show how a liver tumor responds to the chemotherapy given during Transcatheter Arterial Chemoembolization (TACE).

DETAILED DESCRIPTION:
MultiHance is approved by the Food and Drug Administration (FDA) for use as a contrast material for Magnetic Resonance Imaging (MRI) scans of the central nervous system. It is believed that using MultiHance may be able to help doctors tell normal liver cells apart from active tumor and from tumor affected by the chemotherapy. In this way, MultiHance may improve the way patients with hepatocellular carcinoma are managed clinically.

We hypothesize that the Multi-Hance contrast material will provide better image definition of treated liver tumor(s) on MRI imaging in comparison to other commercially available contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between the ages of 18 - 80 seen in the cardiovascular and interventional radiology clinic who are scheduled for TACE.
* International Normalized Ratio (INR) <1.4
* Platelet count > 80,000

Exclusion Criteria:

* Contraindications to TACE procedure
* Unable to have an MRI Scan
* Allergy or hypersensitivity reactions to gadolinium or any other ingredients, including benzyl alcohol
* Patients with sickle cell anemia , hemoglobinopathies and other hemolytic anemias
* Known clinical hypersensitivity or a history of asthma or allergic respiratory disorders
* Patients with advanced renal failure (those currently requiring dialysis or with a Glomerular Filtration Rate<15cc/min)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Kamel, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January, 2008 to May, 2012
  People with hepatocellular carcinoma who were candidates for TACE who were referred to Johns Hopkins Hospital.
Pre-assignment Details: none observed
Groups:
- Gadabenate Dimeglumine( Multihance): If patient did not participate in this study (by signing consent), they could receive any other contrast used routinely at this facility including the contrast used in this study
  gadobenate dimeglumine (MultiHance): The contrast agent, gadobenate dimeglumine, will be used during MRI imaging for both the baseline and 1 month f/u studies.
Period: Overall Study
Arm/Group | Gadabenate Dimeglumine( Multihance)
Started | 45
Completed | 19
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Gadobenate Dimeglumine (Multi Hance)
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] | 60.9 [43 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 33
Region of Enrollment [Count of Participants; unit: Participants] — Percentage of enhancement changes observed using Triple-phase MultiHance-enhanced MRI
  Participants
    United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Nodule Size
Description: Maximal nodule size measured in centimeters
Time Frame: 3 months
Population: The number of participants analyzed reflects the number of participants for whom data was available.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Multihance: If patient did not participate in this study (by signing consent), they could receive any other contrast used routinely at this facility including the contrast used in this study
  gadobenate dimeglumine (MultiHance): The contrast agent, gadobenate dimeglumine, will be used during MR imaging for both the baseline and 1 month f/u studies.
Arm/Group | Multihance
Number analyzed (Participants) | 19
centimeters | 6.4 (4.5)

2. Primary Outcome: Nodule Enhancement
Description: Percent area of nodule with enhancement
Time Frame: 3 month
Population: Number of participants analyzed reflects the number of participants for whom data was available
Measure: Mean (Standard Deviation); unit: percent enhancement
Arm/Group | Multihance
Number analyzed (Participants) | 19
percent enhancement | 32.8 (30.7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Gadobenate Dimeglumine (Multi Hance)
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No